CLINICAL TRIAL: NCT02042365
Title: Prospective Multicentre Study Assessing the Feasibility of Enhanced Recovery After Sleeve Gastrectomy for Obesity
Acronym: SLEEVERAS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHU-0178
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Obesity
Keywords: Enhanced recovery,; sleeve gastrectomy,
MeSH Terms: conditions — Obesity | interventions — Enhanced Recovery After Surgery

GROUPS / COHORTS (1):
- ERAS (Enhanced recovery after surgery): This observational study evaluates the feasibility of ERAS pathway in six French departments of surgery located at Clermont-Ferrand, Bordeaux, Montpellier, Amiens, Strasbourg and Aurillac
  Interventions: Procedure: ERAS (Enhanced recovery after surgery)

INTERVENTIONS:
Procedure: ERAS (Enhanced recovery after surgery)

SUMMARY:
The primary purpose of the study is to test the feasibility of a protocol of enhanced recovery after surgery for reducing the total length of hospital stay in a large scale setting

DETAILED DESCRIPTION:
This observational study evaluates the feasibility of ERAS pathway in six French departments of surgery located at Clermont-Ferrand, Bordeaux, Montpellier, Amiens, Strasbourg and Aurillac.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients undergoing a sleeve gastrectomy Patients having signed the informed consent Patients over 18 year old ASA 1-3 Obesity with indication for surgery according the guidelines of the French High Authority for Health BMI < 50 kg/m2 No contra-indication for general anesthésia

Exclusion Criteria:

contra-indication for general anesthésia Age under 18 years ASA 4 BMI > 50 kg/m2 Patients having other serious comorbidities: cardiac, pulmonary, diabete, immunodepression, coagulopathy ou anticoagulant therapy Pregnancy Patients living alone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients undergoing a sleeve gastrectomy
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | at day 1
  Posoperative day when the patients satisfies the criteria of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Karem SLIM, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France